CLINICAL TRIAL: NCT04405388
Title: Spermidine Anti-Hypertension Study
Acronym: SMARTEST
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Medical University of Graz (Other)
Collaborators: University of Graz (Other); ETH Zurich (Other); Institut National de la Santé Et de la Recherche Médicale, France (Other Government); University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 30-468 ex 17/18
Record Dates: First submitted 2020-02-25; First posted 2020-05-28 (Actual); Last update posted 2023-01-10 (Actual); Status verified 2023-01

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Spermidine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Spermidine first (Other): First treatment period (8 weeks) will be 4 mg spermidine per day orally. Afterwards 4 weeks of wash-out followed by 8 weeks of placebo treatment.
  Interventions: Drug: Placebo; Drug: Spermidine
- Placebo first (Other): First treatment period (8 weeks) will be placebo. Afterwards 4 weeks of wash-out followed by 8 weeks of 4 mg spermidine per day orally.
  Interventions: Drug: Placebo; Drug: Spermidine

INTERVENTIONS:
Drug: Placebo — Placebo will be given orally as capsule (same size and weight as Spermidine capula)
Drug: Spermidine — Spermidine will be given orally as capsule (4mg/day)

SUMMARY:
The impact of daily spermidine application on arterial blood pressure and other secondary parameters will be evaluated in a double-blind single center 46 patients cross-over study.

DETAILED DESCRIPTION:
Arterial hypertension is a central risk factor for cardiovascular disease, major cardiovascular events and mortality. Treatment of arterial hypertension necessitates lifestyle modifications, but often also requires medical intervention. In most cases, a combination of two or more anti-hypertensive drugs is recommended and necessary for reaching the target blood pressure levels.

Hypotheses / research questions/objectives Spermidine potentiates the blood pressure lowering effect of standard anti-hypertensive medications, particularly when a combination of at least two first-line drugs (as recommended by the European Society of Cardiology guidelines) has not resulted in sufficient and adequate blood pressure control.

Approach/methods Spermidine Anti-Hypertension Study (SMARTEST) is a prospective, randomized and double-blind placebo-controlled single-centre trial with a balanced 2x2 crossover design, where 46 medically pre-treated hypertensive patients will be subsequently treated with spermidine and placebo (each for eight weeks) in two arms of opposite treatment sequence. A washout period of four weeks will separate the two intervention periods in both arms.

Patients will undergo physical examination, ECG (electrocardiogram), echocardiography, and blood draws at four time points coinciding with the baseline and termination of each treatment at: 0, 8, 12, and 20 weeks of/after recruitment at the Department of Cardiology, Medical University of Graz. In addition, 24-hour ambulatory blood pressure (24-h BP) monitoring (BPM; Mobil-O-Graph®) and on-site blood pressure will be obtained (the device will be sent back to the hospital the following day) at these time points. A 6-minute walk test (6MWT) will be performed at every visit.

Spermidine will be administered orally as an approved dietary supplement (spermidine-rich wheat germ extract) at a dose of 4 mg spermidine per day for eight weeks. The primary outcome will be arterial systolic blood pressure at 24h BPM. Further secondary outcomes/safety outcomes will be:

24-h BP: analysis of systolic, diastolic and mean arterial blood pressures and pulse wave analysis; on site ambulatory blood pressure; 6 minute walk test distance (difference in meters); laboratory analysis; ECG - standard parameters; Echocardiography: standard parameters as well as strain analysis

ELIGIBILITY:
Inclusion Criteria:

* Able to provide signed and dated informed consent form
* Persistant arterial hypertension with systolic blood pressure above 150 mmHg during hospitalisation and the day of randomisation
* Stable anti-hypertensive medication with at least two guideline-recommended anti-hypertensive drugs

Exclusion Criteria:

* Systolic blood pressure ≥180mmHg on the day of randomisation
* Spermidine intolerance
* Significant renal impairment defined as glomerular filtration rate < 45ml/min
* Insulin-dependent diabetes mellitus (IDDM)
* Wheat allergy or gluten intolerance
* Life expectancy of less than 12 months
* Participation in another clinical trial

Ages: 19 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2020-02-25 (Actual); Primary Completion 2024-11-15 (Estimated); Study Completion 2024-11-15 (Estimated)

PRIMARY OUTCOMES:
Systolic blood pressure in an ambulatory 24h blood pressure measurement | up to 24 weeks
  Patients will get RR recordings in an ambulatory setting

SECONDARY OUTCOMES:
Pulse wave velocity | up to 24 weeks
  recorded with the Mobil-O-Graph® PWA, I.E.M. GmbH, Stolberg, Germany
diastolic blood pressure | up to 24 weeks
  recorded with the Mobil-O-Graph® PWA, I.E.M. GmbH, Stolberg, Germany
mean blood pressure | up to 24 weeks
  recorded with the Mobil-O-Graph® PWA, I.E.M. GmbH, Stolberg, Germany
central blood pressure | up to 24 weeks
  recorded with the Mobil-O-Graph® PWA, I.E.M. GmbH, Stolberg, Germany
6 minute walk test | up to 24 weeks
  tested at every visit

CONTACTS AND LOCATIONS:
Overall Officials: Dirk von Lewinski, MD, Principal Investigator — MUG; Simon Sedej, PhD, Study Director — Medical University of Graz; Tobias Eisenberg, PhD, Study Director — University of Graz; Mahmoud Abdellatif, MD, PhD, Study Director — Medical University of Graz
Locations (1):
- Medical University of Graz, Graz, Austria

IPD SHARING:
Plan to Share IPD: No
individual data will only be shared after approval of the local EC

REFERENCES:
- [Result] Eisenberg T, Abdellatif M, Schroeder S, Primessnig U, Stekovic S, Pendl T, Harger A, Schipke J, Zimmermann A, Schmidt A, Tong M, Ruckenstuhl C, Dammbrueck C, Gross AS, Herbst V, Magnes C, Trausinger G, Narath S, Meinitzer A, Hu Z, Kirsch A, Eller K, Carmona-Gutierrez D, Buttner S, Pietrocola F, Knittelfelder O, Schrepfer E, Rockenfeller P, Simonini C, Rahn A, Horsch M, Moreth K, Beckers J, Fuchs H, Gailus-Durner V, Neff F, Janik D, Rathkolb B, Rozman J, de Angelis MH, Moustafa T, Haemmerle G, Mayr M, Willeit P, von Frieling-Salewsky M, Pieske B, Scorrano L, Pieber T, Pechlaner R, Willeit J, Sigrist SJ, Linke WA, Muhlfeld C, Sadoshima J, Dengjel J, Kiechl S, Kroemer G, Sedej S, Madeo F. Cardioprotection and lifespan extension by the natural polyamine spermidine. Nat Med. 2016 Dec;22(12):1428-1438. doi: 10.1038/nm.4222. Epub 2016 Nov 14. PMID 27841876
- [Result] Wirth M, Benson G, Schwarz C, Kobe T, Grittner U, Schmitz D, Sigrist SJ, Bohlken J, Stekovic S, Madeo F, Floel A. The effect of spermidine on memory performance in older adults at risk for dementia: A randomized controlled trial. Cortex. 2018 Dec;109:181-188. doi: 10.1016/j.cortex.2018.09.014. Epub 2018 Oct 4. PMID 30388439

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-23): https://cdn.clinicaltrials.gov/large-docs/88/NCT04405388/Prot_SAP_000.pdf